CLINICAL TRIAL: NCT00215891
Title: PEG-Interferon a-2b + Ribavirin for Treatment of Chronic Hepatitis C Infection in HIV-Infected Persons Not Previously Treated With Interferon
Brief Title: PEG-Interferon a-2b + Ribavirin for Treatment of Chronic HRN 005 Hepatitis C Infection in HIV-Infected Persons Not Previously Treated With Interferon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hepatitis Resource Network (Other)
Collaborators: Integrated Therapeutics Group (Industry); Subsidiary of Schering-Plough (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRN 005
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Hepatitis C Infection in HIV-Infected Persons; HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Ribavirin

INTERVENTIONS:
Drug: PEG-Interferon a-2b + Ribavirin

SUMMARY:
Objectives:

Primary To compare the sustained virologic response (SVR) of PEGIntron plus ribavirin among patients receiving 48 weeks versus 72 weeks of therapy (defined as undetectable HCV RNA level 24 weeks after discontinuing therapy).

Secondary

* To evaluate the safety and tolerability PEG Intron in combination with ribavirin for treatment of Chronic Hepatitis C (CHC) infection in patients co-infected with Human Immunodeficiency Virus (HIV).
* To determine the early virologic response of patients receiving PEGIntron plus ribavirin at Treatment Week 24

Study Design:

All qualifying patients will enter the treatment phase and be dosed as follows:

Peginterferon a-2b 1.5mg/kg by subcutaneous route once weekly plus

Ribavirin:

* 800 mg (400 mg bid) if body weight < 65 kg
* 1000 mg (400 mg a.m. and 600 mg p.m.) if body weight > 65 kg and < 85 kg
* 1200 mg (600 mg bid) if body weight > 85 kg and < 105 kg
* 1400 mg (600 mg a.m. and 800 mg p.m.) if body weight > 105 kg

At Treatment Week 24, all participants with detectable HCV-RNA will be discontinued from treatment and followed for a Post Treatment period of 24 weeks. Participants with undetectable HCV-RNA values at Treatment Week 24 will be randomized to either:

* Group A: an additional 24 weeks of previously assigned Peginterferon a-2b + Ribavirin therapy, for a total of 48 weeks of treatment.
* Group B: an additional 48 weeks of previously assigned Peginterferon a-2b + Ribavirin therapy, for a total of 72 weeks of treatment.

Study Population:

300 HIV infected adults with chronic hepatitis C infection who have not been treated previously with interferon therapy.

Dosage and Administration:

Peginterferon a-2b 1.5mg/kg by subcutaneous route once weekly plus

Ribavirin:

* 800 mg (400 mg bid) if body weight < 65 kg
* 1000 mg (400 mg a.m. and 600 mg p.m.) if body weight > 65 kg and < 85 kg
* 1200 mg (600 mg bid) if body weight > 85 kg and < 105 kg
* 1400 mg (600 mg a.m. and 800 mg p.m.) if body weight > 105 kg

Efficacy Evaluations:

Laboratory analysis, liver biopsies, quality of life assessments, and changes in Peginterferona-2b and Ribavirin dosages will be obtained.

Safety Evaluations:

* Assessment of laboratory evaluations
* vital signs
* incidence and severity of adverse experiences
* dose adjustments
* premature withdrawal for safety reasons
* progression of disease as measured by HCV viral load
* AIDS defining events

ELIGIBILITY:
Inclusion Criteria:

5.2 Inclusion Criteria

To be eligible for this trial, patients must have documentation of the following:

5.2.1 Written informed consent specific to this protocol obtained prior to screening and willingness to participate in and comply with the study.

5.2.2 Male and female patients >18 years of age.

5.2.3 Detectable plasma HCV-RNA by RT-PCR or other assay (bDNA).

5.2.4 HCV genotype result must be available at screening (historical determinations of genotype are acceptable).

5.2.5 Evidence of HIV infection (reactive HIV antibody with Western blot confirmation).

5.2.6 Compensated liver disease with the following laboratory parameters at screening (results within 1 month of screening):

* Hemoglobin values of ³ 11 gm/dL
* WBC ³ 3,000/mm3
* Neutrophil count ³1,250/mm3
* Platelets ³ 70,000/mm3
* Prothrombin time £ 3 seconds prolonged compared to control, or equivalent INR ratio
* Bilirubin within 20% of the upper limit of normal (unless non-hepatitis related factors such as Gilbert's disease or the use of indinivir explains an indirect bilirubin rise).
* Albumin ³ 3.0 g/dL
* Serum creatinine £ 1.4 mg/dL
* Fasting blood sugar £ 115 mg/dL for non-diabetic patients
* Hemoglobin A1C £ 8.5% for diabetic patients (whether on medication and/or diet controlled)

5.2.7 Thyroid Stimulating Hormone (TSH) within normal limits or thyroid disease under clinical control (within 3 months of screening)

5.2.8 Alpha-fetoprotein (AFP) value within normal limits obtained within the prior year. For patients with results above the upper limit of normal but < 100 ng/mL both of the following are required:

* Alpha-fetoprotein value < 100 ng/mL obtained within 3 months prior to entry AND
* Ultrasound obtained within 3 months prior to entry that is negative for evidence of hepatocellular carcinoma.

5.2.9 CD4 T cell count and HIV RNA level (by RT-PCR) within 1 month of screening:

* CD4 <100 Eligible with HIV RNA <25,000 by RT-PCR
* CD4 > 100 - Eligible with any HIV RNA level by RT-PCR

5.2.10 Stable antiretroviral regimen of FDA-approved agents for at least 4 weeks prior to baseline.

5.2.11 Reconfirmation and documentation that all sexually active female patients of childbearing potential are practicing adequate contraception (intrauterine device, oral contraceptives, progesterone implanted rods [Norplant], medroxyprogesterone acetate [Depo-Provera], surgical sterilization, barrier method [diaphragm + spermicide], or monogamous relationship with a male partner who has had a vasectomy or is using a condom + spermicide) during the treatment period and for 6 months after discontinuation of therapy. Female patients must not breast feed during the treatment period and for 6 months after discontinuation of therapy. A urine pregnancy test obtained at entry prior to the initiation of treatment must be negative.

5.2.12 Reconfirmation and documentation that sexually active male patients are practicing acceptable methods of contraception (vasectomy, use of a condom + spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 6 months after discontinuation of therapy.

5.2.13 Anyone at high risk of coronary artery disease should have a stress test performed prior to entry. This would include, but not be limited to, patients over age 55 who have a history of ischemia or who have a significant history of hypertension, diabetes mellitus, obesity, smoking and/or strong family history of coronary artery disease. Patients with evidence of ischemia on resting or stress EKG, or a history of an arrhythmia, angina or a myocardial infarction within 12 months must be excluded.

5.2.14 Although recommended, liver biopsy is not required for study entry. However, if a liver biopsy has been obtained, within three years of the initial screening visit, the pathology report will be collected with other study data.

Exclusion Criteria:

5.3 Exclusion Criteria

Patients meeting any of the following criteria are not eligible for this trial:

5.3.1 Inability or unwillingness to provide written informed consent specific to this protocol or unwillingness to participate in and comply with the study.

5.3.2 Previous therapy with interferon alfa.

5.3.3 Women with ongoing pregnancy or breast-feeding.

5.3.4 Male partners of women who are pregnant.

5.3.5 Hypersensitivity to interferon or ribavirin.

5.3.6 Evidence of advanced liver disease such as a history of or presence of ascites, bleeding varices, or spontaneous encephalopathy.

5.3.7 Any other causes for chronic liver disease other than chronic hepatitis C.

5.3.8 Hemoglobinopathies (e.g., Thalassemia) or any other cause of hemolytic anemia.

5.3.9 Any known preexisting medical condition that could interfere with a patient's participation in the protocol including: CNS trauma or active seizure disorders requiring medication; poorly controlled diabetes mellitus; serious pulmonary disease; immunologically-mediated diseases; gout; or any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids.

5.3.10 Patients with evidence of ischemia upon stress testing (required for patients at risk of or with a history of coronary artery disease, ECG evidence of ischemia, an arrhythmia, cardiac failure, coronary surgery, uncontrolled hypertension, angina or a myocardial infarction within 12 months).

5.3.11 Active or acute HIV-related opportunistic infection.

5.3.12 Evidence of severe retinopathy (e.g. CMV retinitis, macular degeneration)

5.3.13 History of major organ transplantation with an existing functional graft (including Bone Marrow Transplants)

5.3.14 History of any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) £6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.

5.3.15 Concomitant medication with, rifampin/rifampicin, rifabutin, pyrazinamide, isoniazid, ganciclovir, thalidomide, oxymetholone (Anadrolâ), and immunomodulatory treatments (including supraphysiologic doses of steroids).

5.3.16 Coadministration of didanosine (DDI, dideoxyadenosine 5'-triphosphate) and ribavirin is not recommended.

5.3.17 Evidence of alcohol and/or drug abuse within one year of entry. Patients on methadone programs are not excluded.

5.3.18 Inability to abstain from alcohol throughout the entire course of treatment and follow-up.

5.3.19 History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease.

5.3.20 History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300

PRIMARY OUTCOMES:
Objectives:
Primary
To compare the sustained virologic response (SVR) of PEGIntron plus ribavirin among patients receiving 48 weeks versus 72 weeks of therapy (defined as undetectable HCV RNA level 24 weeks after discontinuing therapy).

SECONDARY OUTCOMES:
Secondary
· To evaluate the safety and tolerability PEG Intron in combination with ribavirin for treatment of Chronic Hepatitis C (CHC) infection in patients co-infected with Human Immunodeficiency Virus (HIV).
· To determine the early virologic response of patients receiving PEGIntron plus ribavirin at Treatment Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sulkowski, MD, Principal Investigator — Hepatitis Resource Network
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States